CLINICAL TRIAL: NCT06444360
Title: Hybrid Type 2 Effectiveness-Implementation Trial of Status Neutral, Integrated Behavioral Activation and Risk Reduction Intervention for Stimulant Use Among Sexually Active Adolescents and Young Adults (Project IMPACT)
Brief Title: Behavioral Activation and Risk Reduction for Stimulant Use Among Sexually Active Adolescents and Young Adults
Acronym: IMPACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Westat (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ATN170; UM2HD111102 (NIH); UM2HD111076 (NIH)
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: HIV
Keywords: Behavioral Activation; risk reduction; intervention; stimulant use; HIV sexual risk reduction
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: The study is a two-arm, multi-site, randomized controlled trial (RCT). IMPACT is a status-neutral intervention that uses behavioral activation (BA)-an evidence-based, cognitive behavior therapy-as a treatment for stimulant use and sexual risk reduction (RR) counseling for adolescents and young adults.
  The IMPACT intervention includes 10 sessions: 2 sessions of HIV sexual risk reduction (RR) counseling, 1 session focused on orienting and rationale of behavioral activation (BA), 6 sessions integrating BA and sexual RR counseling-including pre-exposure prophylaxis (PrEP) or antiretroviral therapy (ART) and HIV care-and 1 final session on strategies for slip-ups and recurrence management.
  The enhanced Standard of Care (eSOC) group includes two HIV sexual RR sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMPACT Group (Experimental): Participants who report stimulant use in the context of condomless sex will be randomized using a 2:1 allocation ratio with two-thirds being allocated to the IMPACT intervention.
  Interventions: Behavioral: IMPACT
- Enhanced Standard of Care (eSOC) Group (Active Comparator): Participants who report stimulant use in the context of condomless sex will be randomized using a 2:1 allocation ratio with one-third being allocated to the eSOC intervention.
  Interventions: Behavioral: eSOC

INTERVENTIONS:
Behavioral: IMPACT — The IMPACT intervention includes 10 sessions: 2 sessions of HIV sexual risk reduction (RR) counseling, 1 session focused on orienting and rationale of behavioral activation (BA), 6 sessions integrating BA and sexual RR counseling (including PrEP or ART and HIV care), and 1 final session on strategies for slip-ups and recurrence management.
  Arms: IMPACT Group
Behavioral: eSOC — The eSOC group includes 2 sessions of HIV sexual RR counseling.
  Arms: Enhanced Standard of Care (eSOC) Group

SUMMARY:
The use of behavioral intervention to reduce stimulant use and concurrent HIV sexual transmission risk.

DETAILED DESCRIPTION:
IMPACT is a Human Immunodeficiency Virus (HIV) status-neutral, behavioral intervention to reduce stimulant use and concurrent HIV sexual transmission risk. This study will evaluate the effectiveness of IMPACT and determine feasibility of implementing IMPACT for translation into real-world practice using a hybrid effectiveness-implementation design.

The IMPACT intervention includes 10 sessions: 2 sessions of HIV sexual risk reduction (RR) counseling, 1 session focused on orienting and rationale of behavioral activation (BA), 6 sessions integrating BA and sexual RR counseling-including pre-exposure prophylaxis (PrEP) or antiretroviral therapy (ART) and HIV care-and 1 final session on strategies for slip-ups and recurrence management.

The enhanced Standard of Care (eSOC) group includes two HIV sexual RR sessions.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-24 years, inclusive, at enrollment
* Male or female
* Self-reports condomless anal or vaginal sex while using stimulants (5 hour prior to, or during sex) within the last 4 months; stimulants is defined as crystal methamphetamine, cocaine, and MDMA (e.g., ecstasy, molly)
* Willing and able to provide written informed consent for study participation
* Access to a computer/smartphone/tablet that can use video chat (e.g., Zoom or Google Meet)
* Provide a mailing address where they can receive a package
* Access to stable internet that they can use for more than 2 hours at a time
* Have a private place (where no one else can see or hear) where they can complete visits online
* Reside within the continental U.S.

Exclusion Criteria:

* Unable to provide informed consent due to severe mental or physical illness
* Concurrent enrollment in another HIV prevention or treatment study (enrollment in a substance treatment program is acceptable)
* Randomized to IMPACT arm prior to March 2025 study stop
* Non-English-speaking
* Is currently incarcerated or pending incarceration
* Is currently pregnant or planning to become pregnant
* Any other medical condition, medical/behavioral intervention, or other condition that, in the opinion of the Project Lead or designee, could interfere with the safety of participants or staff, adherence to study procedures, or compromise interpretation of study results

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Distinct acts of condomless sex without the protection of PrEP or viral suppression. | Participants will recall and report acts of condomless sex and medication adherence for the 30 days prior to each of 4 visits: Baseline, Month 4, Month 8 and Month 12.
  The number of times participants report engaging in condomless sex without the protection of PrEP (for those not living with HIV) or viral suppression (for those living with HIV).

SECONDARY OUTCOMES:
Days of stimulant use | Participants will recall and report the number of days they used stimulants out of the 30 days prior to each of 4 visits and will also have urine drug testing done. The visits are at: Baseline, Month 4, Month 8 and Month 12.
  The number of days participants report having used stimulants

CONTACTS AND LOCATIONS:
Overall Officials: Katie Biello, PhD, MPH, Study Chair — Brown University; Matthew Mimiaga, ScD, MPH, Study Chair — University of California, Los Angeles
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - Brown University, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No